CLINICAL TRIAL: NCT00910988
Title: A Randomized Comparison of the Acute Effects of Olanzapine and Ziprasidone on Whole Body Insulin Sensitivity in Healthy Volunteers
Brief Title: Healthy Volunteers Study of the Effects of Olanzapine and Ziprasidone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 08-0540
Record Dates: First submitted 2009-02-03; First posted 2009-06-01 (Estimated); Results first posted 2014-01-15 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Hyperglycemia; Hyperlipidemia
Keywords: healthy; sedentary; men; acute effects of antipsychotic; blood sugar; insulin sensitivity
MeSH Terms: conditions — Hyperglycemia; Hyperlipidemias; Sedentary Behavior; Multiple Endocrine Neoplasia Type 1; Insulin Resistance | interventions — Olanzapine; ziprasidone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- olanzapine (Active Comparator): olanzapine injection in healthy control
  Interventions: Drug: Olanzapine
- ziprasidone (Active Comparator): ziprasidone injection in healthy control
  Interventions: Drug: Ziprasidone
- saline (Placebo Comparator): saline injection in healthy control
  Interventions: Drug: Olanzapine; Drug: Ziprasidone

INTERVENTIONS:
Drug: Olanzapine — olanzapine/Zyprexa
  Other Names: Zyprexa
  Arms: olanzapine; saline
Drug: Ziprasidone — ziprasidone/Geodon
  Other Names: Geodon
  Arms: saline; ziprasidone

SUMMARY:
Primary Aim: To test the acute effects of olanzapine or ziprasidone administration, in comparison to placebo, on insulin sensitivity in antipsychotic-naïve healthy young men, measured as whole-body dextrose infusion rates (mg/kg/min), hepatic glucose production (glucose rate of appearance [Ra]), primarily muscle glucose utilization (glucose rate of disappearance [Rd]), and adipose tissue related free fatty acid production (glycerol rate of appearance [Ra]).

We hypothesize that olanzapine, but not ziprasidone, will result in acute decreases in insulin sensitivity.

Secondary Aim: To test the acute effects of olanzapine or ziprasidone on insulin signaling pathways in antipsychotic naïve healthy young men.

We hypothesize that olanzapine, but not ziprasidone, will result in acute alterations in insulin signaling.

DETAILED DESCRIPTION:
See brief description

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18-45 years
* BMI approximately ≥ 25 and < 35
* insulin approximately ≥ 15 µU/ml or triglyceride approximately ≥ 130 mg/dl

Exclusion Criteria:

* Any DSM-IV Axis I diagnosis
* prisoners
* any serious medical disorder (i.e. metabolic diseases, type 1 or 2 diabetes mellitus, endocrine disease, coagulopathy, clinically significant anemia, acute infection)
* taking prescription medications
* non-sedentary lifestyle with > 3 hours of exercise per week

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2009-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W Newcomer, MD, Principal Investigator — Washington University School of Medicine and Florida Atlantic University; Ginger Nicol, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Olanzapine (Drug First): Subjects from this group received an olanzapine injection at the first clamp followed by a saline injection at the second clamp.
- Ziprasidone (Drug First): Subjects from this group received a ziprasidone injection at the first clamp followed by a saline injection at the second clamp.
- Olanzapine (Placebo First): Subjects from this group received a saline injection at the first clamp followed by an olanzapine injection at the second clamp.
- Ziprasidone (Placebo First): Subjects from this group received a saline injection at the first clamp followed by a ziprasidone injection at the second clamp.
Period: Overall Study
Arm/Group | Olanzapine (Drug First) | Ziprasidone (Drug First) | Olanzapine (Placebo First) | Ziprasidone (Placebo First)
Started | 16 | 16 | 8 | 6
Completed | 14 | 12 | 5 | 6
Not Completed | 2 | 4 | 3 | 0
Not completed — Lost to Follow-up | 2 | 4 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine (Drug First) | Ziprasidone (Drug First) | Olanzapine (Placebo First) | Ziprasidone (Placebo First) | Total
Number analyzed (Participants) | 16 | 16 | 8 | 6 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] — Intent-To-Treat (eg, completed at least one clamp)
  years | 34.9 (8.9) | 33.2 (8.7) | 31.9 (8.7) | 29.7 (8.7) | 33.1 (8.6)
Age, Continuous [Mean (Standard Deviation); unit: years] — Completer Sample (eg, completed both clamps)
  years | 34.5 (9.1) | 32.9 (9.0) | 37.0 (5.6) | 29.7 (8.7) | 33.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Intent-To-Treat (eg, completed at least one clamp)
  Participants
    Female | 0 | 0 | 0 | 0 | 0
    Male | 16 | 16 | 8 | 6 | 46
Sex/Gender, Customized [Number; unit: participants] — Completer Sample (eg, completed both clamps), which includes 37 subjects
  participants
    Female | 0 | 0 | 0 | 0 | 0
    Male | 14 | 12 | 5 | 6 | 37
Race/Ethnicity, Customized [Number; unit: participants] — Completer Sample (eg, completed both clamps), which includes 37 subjects
  participants
    Caucasian | 5 | 5 | 1 | 4 | 15
    African American | 7 | 5 | 4 | 2 | 18
    Asian | 1 | 0 | 0 | 0 | 1
    Native American | 1 | 1 | 0 | 0 | 2
    Other | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants] — Intent-To-Treat (eg, completed at least one clamp)
  participants
    Caucasian | 5 | 7 | 1 | 4 | 17
    African American | 9 | 6 | 7 | 2 | 24
    Asian | 1 | 1 | 0 | 0 | 2
    Native American | 1 | 1 | 0 | 0 | 2
    Other | 0 | 1 | 0 | 0 | 1
Weight [Mean (Standard Deviation); unit: kilograms] — Intent-To-Treat (eg, completed at least one clamp)
  kilograms | 93.7 (10.5) | 97.4 (15.1) | 114.1 (10.0) | 96.2 (6.0) | 98.9 (13.6)
Weight [Mean (Standard Deviation); unit: kilograms] — Completer Sample (eg, completed both clamps)
  kilograms | 94.6 (10.9) | 96.7 (10.7) | 113.1 (9.4) | 96.2 (6.0) | 98.0 (11.4)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Intent-To-Treat (eg, completed at least one clamp)
  kg/m^2 | 29.49 (2.02) | 30.85 (3.34) | 33.83 (1.90) | 30.84 (1.45) | 30.89 (2.85)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Completer Sample (eg, completed both clamps)
  kg/m^2 | 29.60 (2.13) | 30.86 (2.82) | 33.18 (1.56) | 30.84 (1.45) | 30.69 (2.44)
Waist Circumference [Mean (Standard Deviation); unit: centimeters] — Intent-To-Treat (eg, completed at least one clamp)
  centimeters | 101.5 (8.0) | 103.9 (11.8) | 112.5 (5.0) | 106.2 (8.7) | 104.9 (9.7)
Waist Circumference [Mean (Standard Deviation); unit: centimeters] — Completer Sample (eg, completed both clamps)
  centimeters | 102.0 (8.3) | 104.3 (10.7) | 111.4 (4.2) | 106.2 (8.7) | 104.7 (9.0)
DEXA Total Fat [Mean (Standard Deviation); unit: kilograms] — Intent-To-Treat (eg, completed at least one clamp)
  kilograms | 25.3 (7.0) | 27.4 (8.3) | 32.2 (5.9) | 27.8 (5.5) | 27.6 (7.3)
DEXA Total Fat [Mean (Standard Deviation); unit: kilograms] — Completer Sample (eg, completed both clamps)
  kilograms | 25.8 (7.3) | 26.9 (7.4) | 30.4 (6.9) | 27.8 (5.5) | 27.1 (6.9)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Intent-To-Treat (eg, completed at least one clamp)
  mmHg | 130 (9) | 127 (9) | 135 (14) | 130 (10) | 130 (10)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Completer Sample (eg, completed both clamps)
  mmHg | 130 (10) | 130 (7) | 134 (17) | 130 (10) | 131 (10)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Intent-To-Treat (eg, completed at least one clamp)
  mmHg | 78 (9) | 74 (11) | 81 (13) | 71 (10) | 76 (11)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Completer Sample (eg, completed both clamps)
  mmHg | 80 (8) | 77 (6) | 82 (15) | 71 (10) | 78 (9)
Heart Rate [Mean (Standard Deviation); unit: beats per minute] — Intent-To-Treat (eg, completed at least one clamp)
  beats per minute | 66 (11) | 70 (11) | 62 (9) | 66 (7) | 67 (11)
Heart Rate [Mean (Standard Deviation); unit: beats per minute] — Completer Sample (eg, completed both clamps)
  beats per minute | 67 (12) | 71 (11) | 57 (5) | 66 (7) | 67 (11)
Fasting Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Intent-To-Treat (eg, completed at least one clamp)
  mg/dL | 193.6 (40.3) | 171.9 (37.7) | 171.6 (32.1) | 175.3 (24.2) | 179.8 (36.6)
Fasting Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Completer Sample (eg, completed both clamps)
  mg/dL | 191.9 (41.4) | 169.6 (37.6) | 176.8 (38.4) | 175.3 (24.2) | 179.9 (37.3)
Fasting HDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Intent-To-Treat (eg, completed at least one clamp)
  mg/dL | 41.1 (16.3) | 38.9 (9.0) | 40.5 (10.5) | 29.2 (6.5) | 38.7 (12.3)
Fasting HDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Completer Sample (eg, completed both clamps)
  mg/dL | 42.3 (17.1) | 38.9 (9.6) | 43.4 (11.1) | 29.2 (6.5) | 39.2 (13.3)
Fasting Triglycerides [Mean (Standard Deviation); unit: mg/dL] — Intent-To-Treat (eg, completed at least one clamp)
  mg/dL | 152.8 (52.4) | 125.9 (58.7) | 121.2 (64.0) | 171.0 (55.2) | 140.3 (57.9)
Fasting Triglycerides [Mean (Standard Deviation); unit: mg/dL] — Completer Sample (eg, completed both clamps)
  mg/dL | 152.8 (55.5) | 122.0 (62.1) | 128.6 (79.3) | 171.0 (55.2) | 142.5 (61.3)
Fasting LDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Intent-To-Treat (eg, completed at least one clamp)
  mg/dL | 120.1 (33.2) | 106.7 (28.0) | 104.1 (30.4) | 116.3 (27.2) | 112.2 (30.0)
Fasting LDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Completer Sample (eg, completed both clamps)
  mg/dL | 117.9 (33.5) | 105.2 (26.3) | 104.2 (38.5) | 116.3 (27.2) | 111.6 (30.4)
Fasting Insulin [Mean (Standard Deviation); unit: uIU/mL] — Intent-To-Treat (eg, completed at least one clamp)
  uIU/mL | 16.3 (10.8) | 13.4 (5.1) | 21.1 (7.6) | 17.0 (10.4) | 16.2 (8.7)
Fasting Insulin [Mean (Standard Deviation); unit: uIU/mL] — Completer Sample (eg, completed both clamps)
  uIU/mL | 16.6 (11.5) | 13.6 (5.5) | 20.0 (9.5) | 17.0 (10.4) | 16.2 (9.3)

OUTCOME MEASURES:

1. Primary Outcome: Whole Body Insulin Sensitivity
Description: To evaluate, using a within-subject placebo-controlled comparison, the acute effects of olanzapine or ziprasidone administration on insulin sensitivity in antipsychotic-naïve healthy young men, measured as whole-body dextrose infusion rates (mg/kg/min).
Time Frame: approximately 3 hours
Population: The analysis was per protocol and involved subjects who completed both a clamp that involved an injection of either olanzapine or ziprasidone, and a clamp that involved a placebo injection. Nine subjects did not complete a second clamp as they were lost to follow-up. This resulted in the analysis of 37 participants.
Measure: Mean (Standard Deviation); unit: mg/kg/min
Groups:
- Olanzapine (Drug/Placebo)-Drug: Subjects from this group received olanzapine (10 mg per IM injection) and will receive normal saline at the next visit.
- Olanzapine (Drug/Placebo)-Placebo: Subjects from this group received 0.9% normal saline (1 ml per IM injection) while having received olanzapine at the previous visit.
- Olanzapine (Placebo/Drug)-Placebo: Subjects from this group received 0.9% normal saline (1 ml per IM injection) and will receive olanzapine at the next visit.
- Olanzapine (Placebo/Drug)-Drug: Subjects from this group received olanzapine (10 mg per IM injection) while having received normal saline at previous visit.
- Ziprasidone (Placebo/Drug)-Placebo: Subjects from this group received 0.9% normal saline (1 ml per IM injection) and will receive ziprasidone at the next visit.
- Ziprasidone (Placebo/Drug)-Drug: Subjects from this group received ziprasidone (20 mg per IM injection) while having received normal saline at previous visit.
- Ziprasidone (Drug/Placebo)-Drug: Subjects from this group received ziprasidone (20 mg per IM injection) and will receive normal saline at the next visit.
- Ziprasidone (Drug/Placebo)-Placebo: Subjects from this group received 0.9% normal saline (1 ml per IM injection) while having received ziprasidone at the previous visit.
Arm/Group | Olanzapine (Drug/Placebo)-Drug | Olanzapine (Drug/Placebo)-Placebo | Olanzapine (Placebo/Drug)-Placebo | Olanzapine (Placebo/Drug)-Drug | Ziprasidone (Placebo/Drug)-Placebo | Ziprasidone (Placebo/Drug)-Drug | Ziprasidone (Drug/Placebo)-Drug | Ziprasidone (Drug/Placebo)-Placebo
Number analyzed (Participants) | 14 | 14 | 5 | 5 | 6 | 6 | 12 | 12
mg/kg/min | 4.9 (2.2) | 5.4 (2.6) | 4.1 (1.2) | 2.9 (1.0) | 5.8 (2.2) | 4.7 (1.8) | 4.5 (3.1) | 5.3 (3.3)
Statistical Analysis 1: Comparison: Olanzapine (Drug/Placebo)-Drug vs Olanzapine (Drug/Placebo)-Placebo vs Olanzapine (Placebo/Drug)-Placebo vs Olanzapine (Placebo/Drug)-Drug vs Ziprasidone (Placebo/Drug)-Placebo vs Ziprasidone (Placebo/Drug)-Drug vs Ziprasidone (Drug/Placebo)-Drug vs Ziprasidone (Drug/Placebo)-Placebo; The hypothesis being tested is whether there is a significant effect of one or both antipsychotics on whole body insulin sensitivity. Sample size was calculated using power calculations to detect significant effects of treatment on insulin sensitivity. Drug assignment is a 2-level fixed factor (olanzapine vs ziprasidone) as is order (drug first vs placebo first). Baseline of the dependent variable as well as baseline DEXA total fat were entered into the model as covariates; Test type: Superiority or Other; p = 0.001, ANCOVA — This p-value corresponds to the two way interaction between time and order and is not adjusted for multiple comparisons. The a priori threshold for statistical significance is alpha equal to 0.05. There was no 3 way interaction; Repeated measures ANCOVA with time as the repeated measure, drug assignment as a fixed factor, and order as a fixed factor

2. Primary Outcome: Hepatic Insulin Sensitivity
Description: To evaluate, using a within-subject placebo-controlled comparison, the acute effects of olanzapine or ziprasidone administration on insulin sensitivity in antipsychotic-naïve healthy young men, measured as hepatic glucose production (glucose rate of appearance [Ra]).
Time Frame: approximately 3 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change from basal to insulin phase
Groups:
- Olanzapine, to be Followed by Normal Saline: Subjects from this group received olanzapine (10 mg per IM injection) and will receive normal saline at the next visit.
- Normal Saline, Following Olanzapine: Subjects from this group received 0.9% normal saline (1 ml per IM injection) while having received olanzapine at the previous visit.
- Normal Saline, to be Followed by Olanzapine: Subjects from this group received 0.9% normal saline (1 ml per IM injection) and will receive olanzapine at the next visit.
- Olanzapine, Following Normal Saline: Subjects from this group received olanzapine (10 mg per IM injection) while having received normal saline at previous visit.
- Normal Saline, to be Followed by Ziprasidone: Subjects from this group received 0.9% normal saline (1 ml per IM injection) and will receive ziprasidone at the next visit.
- Ziprasidone, Following Normal Saline: Subjects from this group received ziprasidone (20 mg per IM injection) while having received normal saline at previous visit.
- Ziprasidone, to be Followed by Normal Saline: Subjects from this group received ziprasidone (20 mg per IM injection) and will receive normal saline at the next visit.
- Normal Saline, Following Ziprasidone: Subjects from this group received 0.9% normal saline (1 ml per IM injection) while having received ziprasidone at the previous visit.
Arm/Group | Olanzapine, to be Followed by Normal Saline | Normal Saline, Following Olanzapine | Normal Saline, to be Followed by Olanzapine | Olanzapine, Following Normal Saline | Normal Saline, to be Followed by Ziprasidone | Ziprasidone, Following Normal Saline | Ziprasidone, to be Followed by Normal Saline | Normal Saline, Following Ziprasidone
Number analyzed (Participants) | 14 | 14 | 5 | 5 | 6 | 6 | 12 | 12
% change from basal to insulin phase | 81.0 (9.4) | 79.1 (6.1) | 73.1 (16.2) | 78.5 (8.1) | 84.0 (13.5) | 80.7 (8.5) | 82.1 (8.6) | 83.4 (6.8)

3. Primary Outcome: Peripheral Insulin Sensitivity
Description: To evaluate, using a within-subject placebo-controlled comparison, the acute effects of olanzapine or ziprasidone administration on insulin sensitivity in antipsychotic-naïve healthy young men, measured as primarily muscle glucose utilization (glucose rate of disappearance [Rd]).
Time Frame: approximately 3 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change from basal to insulin phase
Arm/Group | Olanzapine, to be Followed by Normal Saline | Normal Saline, Following Olanzapine | Normal Saline, to be Followed by Olanzapine | Olanzapine, Following Normal Saline | Normal Saline, to be Followed by Ziprasidone | Ziprasidone, Following Normal Saline | Ziprasidone, to be Followed by Normal Saline | Normal Saline, Following Ziprasidone
Number analyzed (Participants) | 14 | 14 | 5 | 5 | 6 | 6 | 12 | 12
% change from basal to insulin phase | 152.2 (88.0) | 183.5 (130.7) | 157.0 (72.2) | 83.7 (60.5) | 208.2 (96.0) | 161.0 (85.0) | 135.6 (128.4) | 185.3 (136.5)

4. Primary Outcome: Adipose Tissue Insulin Sensitivity
Description: To evaluate, using a within-subject placebo-controlled comparison, the acute effects of olanzapine or ziprasidone administration on insulin sensitivity in antipsychotic-naïve healthy young men, measured as free fatty acid release (glycerol rate of appearance [Ra]).
Time Frame: approximately 3 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change from basal to insulin phase
Arm/Group | Olanzapine, to be Followed by Normal Saline | Normal Saline, Following Olanzapine | Normal Saline, to be Followed by Olanzapine | Olanzapine, Following Normal Saline | Normal Saline, to be Followed by Ziprasidone | Ziprasidone, Following Normal Saline | Ziprasidone, to be Followed by Normal Saline | Normal Saline, Following Ziprasidone
Number analyzed (Participants) | 14 | 14 | 5 | 5 | 6 | 6 | 12 | 12
% change from basal to insulin phase | 43.3 (13.2) | 45.2 (15.8) | 52.8 (13.8) | 53.1 (14.4) | 39.5 (14.6) | 37.6 (8.9) | 47.8 (11.7) | 44.4 (12.1)
Statistical Analysis 1: Comparison: Olanzapine, to be Followed by Normal Saline vs Normal Saline, Following Olanzapine vs Normal Saline, to be Followed by Olanzapine; The null hypothesis is that olanzapine and ziprasidone would result in acute decreases in insulin sensitivity compared to placebo at adipose tissue, which was measured by evaluating the rate of appearance of labeled glycerol. The alternative hypothesis is that olanzapine, but not ziprasidone, would result in acute decreases in insulin sensitivity compared to placebo at adipose tissue; Test type: Superiority or Other; p = 0.57, ANCOVA — This p-value corresponds to the 3 way interaction between time, drug (olanzapine vs ziprasidone), and order (drug first vs placebo first) and is not adjusted for multiple comparisons

ADVERSE EVENTS:
Arm/Group | Olanzapine, to be Followed by Normal Saline | Normal Saline, Following Olanzapine | Normal Saline, to be Followed by Olanzapine | Olanzapine, Following Normal Saline | Normal Saline, to be Followed by Ziprasidone | Ziprasidone, Following Normal Saline | Ziprasidone, to be Followed by Normal Saline | Normal Saline, Following Ziprasidone
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 12 | 12 | 63 | 82 | 72 | 88 | 12 | 10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Olanzapine, to be Followed by Normal Saline | Normal Saline, Following Olanzapine | Normal Saline, to be Followed by Olanzapine | Olanzapine, Following Normal Saline | Normal Saline, to be Followed by Ziprasidone | Ziprasidone, Following Normal Saline | Ziprasidone, to be Followed by Normal Saline | Normal Saline, Following Ziprasidone
Itching, rash, or hives-during past week (General disorders) | 0/14 | 1/14 | 0/5 | 0/5 | 0/6 | 1/6 | 1/12 | 1/12 — Any report of itching, rash, or hives anytime during the past 7 days.
Chest pain-during past week (General disorders) | 0/14 | 0/14 | 0/5 | 1/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of chest pain anytime during the past 7 days.
Heart palpitations-during past week (General disorders) | 0/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 1/12 | 0/12 — Any report of heart palpitations anytime during the past 7 days.
Dizziness-during past week (General disorders) | 0/14 | 0/14 | 0/5 | 1/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of dizziness anytime during the past 7 days.
Dizziness-30 minutes post injection (General disorders) | 1/14 | 1/14 | 0/5 | 0/5 | 0/6 | 0/6 | 1/12 | 0/12 — Any report of dizziness 30 minutes following an injection of antipsychotic or saline.
Dizziness-1 hour post meal (Gastrointestinal disorders) | 0/14 | 1/14 | 0/5 | 0/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of dizziness 1 hour following the meal (after the clamp procedure).
Dizziness-prior to discharge (General disorders) | 1/6 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of dizziness prior to discharge from the hospital.
Angry or agitated-during past week (General disorders) | 1/14 | 1/14 | 1/5 | 0/5 | 2/6 | 0/6 | 0/12 | 0/12 — Any report of being angry or agitated anytime during the past 7 days.
Angry or agitated-prior to injection (General disorders) | 0/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 1/12 | 0/12 — Any report of being angry or agitated prior to injection of antipsychotic or saline.
Angry or agitated-end of clamp (General disorders) | 0/14 | 0/14 | 0/5 | 2/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of being angry or agitated at the end of the clamp procedure.
Confused-30 minutes post injection (General disorders) | 1/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of confusion 30 minutes following an injection of antipsychotic or saline.
Confused-end of clamp (General disorders) | 0/14 | 0/14 | 0/5 | 1/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of confusion at the end of the clamp procedure.
Headache-during past week (General disorders) | 3/14 | 3/14 | 3/5 | 2/5 | 0/6 | 0/6 | 1/12 | 1/12 — Any report of headache anytime during the past 7 days.
Headache-prior to injection (General disorders) | 1/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of headache prior to injection of antipsychotic or saline.
Headache-30 minutes post injection (General disorders) | 2/14 | 0/14 | 1/5 | 1/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of headache 30 minutes following an injection of antipsychotic or saline.
Headache-end of clamp (General disorders) | 0/14 | 1/14 | 0/5 | 0/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of headache at the end of the clamp procedure.
Sad, blue, or depressed-during past week (General disorders) | 1/14 | 0/14 | 0/5 | 0/5 | 1/6 | 0/6 | 0/12 | 0/12 — Any report of sadness, feeling blue, or feeling depressed anytime during the past 7 days .
Worried, anxious-during past week (General disorders) | 4/14 | 3/14 | 1/5 | 0/5 | 1/6 | 1/6 | 2/12 | 1/12 — Any report of being worried or anxious anytime during the past 7 days .
Worried, anxious-prior to injection (General disorders) | 3/14 | 2/14 | 1/5 | 0/5 | 2/6 | 0/6 | 3/12 | 1/12 — Any report of being worried or anxious prior to injection of antipsychotic or saline.
Worried, anxious-30 minutes post injection (General disorders) | 1/14 | 0/14 | 0/5 | 0/5 | 1/6 | 0/6 | 0/12 | 0/12 — Any report of being worried or anxious 30 minutes following an injection of antipsychotic or saline.
Worried, anxious-end of clamp (General disorders) | 0/14 | 0/14 | 0/5 | 2/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of being worried or anxious at the end of the clamp procedure.
Tiredness, fatigue-during past week (General disorders) | 5/14 | 4/14 | 2/5 | 2/5 | 3/6 | 4/6 | 4/12 | 6/12 — Any report of being tired or fatigued anytime during the past 7 days .
Tiredness, fatigue-prior to injection (General disorders) | 5/14 | 3/14 | 2/5 | 3/5 | 3/6 | 3/6 | 5/12 | 5/12 — Any report of being tired or fatigued prior to injection of antipsychotic or saline.
Tiredness, fatigue-30 minutes post injection (General disorders) | 9/14 | 3/14 | 1/5 | 1/5 | 3/6 | 4/6 | 6/12 | 7/12 — Any report of being tired or fatigued 30 minutes following an injection of antipsychotic or saline.
Tiredness, fatigue-end of clamp (General disorders) | 9/14 | 3/14 | 2/5 | 3/5 | 2/6 | 4/6 | 10/12 | 5/12 — Any report of being tired or fatigued at the end of the clamp procedure.
Tiredness, fatigue-1 hour post meal (General disorders) | 8/14 | 1/14 | 0/5 | 3/5 | 1/6 | 3/6 | 9/12 | 3/12 — Any report of being tired or fatigued 1 hour following the meal (after the clamp procedure).
Tiredness, fatigue-prior to discharge (General disorders) | 5/7 | 0/14 | 0/5 | 2/3 | 0/6 | 0/6 | 2/5 | 0/12 — Any report of being tired or fatigued prior to discharge from the hospital.
Dry mouth, thirsty-during past week (General disorders) | 2/14 | 1/14 | 0/5 | 0/5 | 0/6 | 0/6 | 1/12 | 0/12 — Any report of dry mouth or thirstiness anytime during the past 7 days .
Dry mouth, thirsty-prior to injection (General disorders) | 2/14 | 1/14 | 0/5 | 0/5 | 1/6 | 0/6 | 3/12 | 0/12 — Any report of dry mouth or thirstiness prior to injection of antipsychotic or saline .
Dry mouth, thirsty-30 minutes post injection (General disorders) | 3/14 | 2/14 | 0/5 | 1/5 | 2/6 | 2/6 | 4/12 | 3/12 — Any report of dry mouth or thirstiness 30 minutes following an injection of antipsychotic or saline.
Dry mouth, thirsty-end of clamp (General disorders) | 1/14 | 2/14 | 0/5 | 0/5 | 0/6 | 0/6 | 2/12 | 0/12 — Any report of dry mouth or thirstiness at the end of the clamp procedure.
Dry mouth, thirsty-1 hour post meal (General disorders) | 1/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 1/12 | 0/12 — Any report of dry mouth or thirstiness 1 hour following the meal (after the clamp procedure).
Extra saliva-during past week (General disorders) | 0/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 1/12 | 1/12 — Any report of extra saliva anytime during the past 7 days.
Constipation, diarrhea-during past week (General disorders) | 0/14 | 1/14 | 0/5 | 0/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of constipation or diarrhea anytime during the past 7 days.
Fever-during past week (General disorders) | 0/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 1/12 | 0/12 — Any report of fever anytime during the past 7 days.
Hypotension-end of clamp (General disorders) | 4/14 | 0/14 | 0/5 | 1/5 | 0/6 | 1/6 | 5/12 | 0/12 — Any report of hypotension at the end of the clamp procedure.
Hypotension-1 hour post meal (General disorders) | 1/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of hypotension 1 hour following the meal (after the clamp procedure).
Drowsiness, somnolence-during past week (General disorders) | 5/14 | 4/14 | 2/5 | 2/5 | 2/6 | 4/6 | 3/12 | 6/12 — Any report of drowsiness or somnolence anytime during the past 7 days .
Drowsiness, somnolence-prior to injection (General disorders) | 5/14 | 6/14 | 2/5 | 4/5 | 3/6 | 3/6 | 4/12 | 5/12 — Any report of drowsiness or somnolence prior to injection of antipsychotic or saline.
Drowsiness, somnolence-30 minutes post injection (General disorders) | 12/14 | 5/14 | 2/5 | 4/5 | 3/6 | 6/6 | 8/12 | 6/12 — Any report of drowsiness or somnolence 30 minutes following an injection of antipsychotic or saline.
Drowsiness, somnolence-end of clamp (General disorders) | 11/14 | 3/14 | 3/5 | 5/5 | 1/6 | 6/6 | 12/12 | 2/12 — Any report of drowsiness or somnolence at the end of the clamp procedure.
Drowsiness, somnolence-1 hour post meal (General disorders) | 12/14 | 0/14 | 0/5 | 4/5 | 1/6 | 3/6 | 9/12 | 0/12 — Any report of drowsiness or somnolence 1 hour following the meal (after the clamp procedure).
Drowsiness, somnolence-prior to discharge (General disorders) | 4/9 | 0/14 | 0/5 | 2/3 | 0/6 | 1/1 | 2/5 | 0/12 — Any report of drowsiness or somnolence prior to discharge from the hospital.
Stiff muscles or jaw-during past week (General disorders) | 2/14 | 1/14 | 0/5 | 0/5 | 0/6 | 1/6 | 1/12 | 1/12 — Any report of stiff muscles or jaw anytime during the past 7 days.
Stiff muscles or jaw-30 minutes post injection (General disorders) | 1/14 | 2/14 | 1/5 | 0/5 | 0/6 | 1/6 | 0/12 | 1/12 — Any report of stiff muscles or jaw 30 minutes following an injection of antipsychotic or saline.
Stiff muscles or jaw-end of clamp (General disorders) | 1/14 | 2/14 | 2/5 | 0/5 | 0/6 | 0/6 | 0/12 | 1/12 — Any report of stiff muscles or jaw at the end of the clamp procedure.
Stiff muscles or jaw-1 hour post meal (General disorders) | 1/14 | 1/14 | 0/5 | 0/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of stiff muscles or jaw 1 hour following the meal (after the clamp procedure).
Muscle tenderness-during past week (General disorders) | 1/14 | 2/14 | 0/5 | 0/5 | 0/6 | 0/6 | 1/12 | 0/12 — Any report of muscle tenderness anytime during the past 7 days.
Muscle tenderness-30 minutes post injection (General disorders) | 1/14 | 1/14 | 0/5 | 0/5 | 1/6 | 1/6 | 1/12 | 0/12 — Any report of muscle tenderness 30 minutes following an injection of antipsychotic or saline.
Muscle tenderness-1 hour post meal (General disorders) | 0/14 | 0/14 | 1/5 | 1/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of muscle tenderness 1 hour following the meal (after the clamp procedure).
Big appetite-during past week (General disorders) | 8/14 | 6/14 | 5/5 | 4/5 | 5/6 | 3/6 | 9/12 | 7/12 — Any report of a big appetite anytime during the past 7 days.
Trouble sleeping-during past week (General disorders) | 6/14 | 3/14 | 2/5 | 1/5 | 5/6 | 6/6 | 5/12 | 4/12 — Any report of trouble sleeping anytime during the past 7 days.
Heartburn-during past week (General disorders) | 2/14 | 3/14 | 2/5 | 2/5 | 0/6 | 1/6 | 2/12 | 3/12 — Any report of heartburn anytime during the past 7 days.
Shakiness-during past week (General disorders) | 1/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 1/12 | 0/12 — Any report of shakiness anytime during the past 7 days.
Involuntary movements-during past week (General disorders) | 0/14 | 0/14 | 1/5 | 0/5 | 1/6 | 0/6 | 1/12 | 0/12 — Any report of involuntary movements anytime during the past 7 days.
Involuntary movements-30 minutes post injection (General disorders) | 0/14 | 0/14 | 1/5 | 0/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of involuntary movements 30 minutes following an injection of antipsychotic or saline.
Involuntary movements-end of clamp (General disorders) | 1/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of involuntary movements at the end of the clamp procedure.
Restlessness-during past week (General disorders) | 2/14 | 0/14 | 0/5 | 0/5 | 1/6 | 1/6 | 1/12 | 0/12 — Any report of restlessness anytime during the past 7 days.
Restlessness-prior to injection (General disorders) | 3/14 | 2/14 | 0/5 | 0/5 | 0/6 | 0/6 | 1/12 | 1/12 — Any report of restlessness prior to injection of antipsychotic or saline.
Restlessness-30 minutes post injection (General disorders) | 4/14 | 1/14 | 1/5 | 1/5 | 2/6 | 2/6 | 2/12 | 0/12 — Any report of restlessness 30 minutes following an injection of antipsychotic or saline.
Restlessness-end of clamp (General disorders) | 9/14 | 3/14 | 1/5 | 2/5 | 1/6 | 1/6 | 2/12 | 2/12 — Any report of restlessness at the end of the clamp procedure.
Restlessness-1 hour post meal (General disorders) | 2/14 | 0/14 | 0/5 | 1/5 | 0/6 | 0/6 | 2/12 | 1/12 — Any report of restlessness 1 hour following the meal (after the clamp procedure).
Restlessness-prior to discharge (General disorders) | 0/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 1/3 | 0/12 — Any report of restlessness prior to discharge from the hospital.
Runny nose-during past week (General disorders) | 0/14 | 1/14 | 1/5 | 1/5 | 1/6 | 0/6 | 2/12 | 0/12 — Any report of a runny nose anytime during the past 7 days.
Runny nose-prior to injection (General disorders) | 0/14 | 0/14 | 1/5 | 0/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of a runny nose prior to injection of antipsychotic or saline.
Runny nose-30 minutes post injection (General disorders) | 0/14 | 0/14 | 0/5 | 0/5 | 0/6 | 1/6 | 0/12 | 0/12 — Any report of a runny nose 30 minutes following an injection of antipsychotic or saline.
Runny nose-end of clamp (General disorders) | 0/14 | 1/14 | 0/5 | 0/5 | 0/6 | 1/6 | 0/12 | 0/12 — Any report of a runny nose at the end of the clamp procedure.
Tremor-during past week (General disorders) | 1/14 | 1/14 | 1/5 | 1/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of tremors anytime during the past 7 days.
Tremor-1 hour post meal (General disorders) | 1/14 | 1/14 | 0/5 | 0/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of tremors 1 hour following the meal (after the clamp procedure).
Nausea-during past week (General disorders) | 1/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 1/12 | 0/12 — Any report of nausea anytime during the past 7 days.
Nausea-prior to injection (General disorders) | 0/14 | 1/14 | 0/5 | 0/5 | 1/6 | 0/6 | 0/12 | 0/12 — Any report of nausea prior to injection of antipsychotic or saline.
Nausea-end of clamp (General disorders) | 0/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 1/12 | 0/12 — Any report of nausea at the end of the clamp procedure.
Vomiting-during past week (General disorders) | 0/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 1/12 | 0/12 — Any report of vomiting anytime during the past 7 days.
Weakness-30 minutes post injection (General disorders) | 1/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 1/12 | 0/12 — Any report of weakness 30 minutes following an injection of antipsychotic or saline.
Weakness-end of clamp (General disorders) | 0/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 1/12 | 0/12 — Any report of weakness at the end of the clamp procedure.
Weakness-1 hour post meal (General disorders) | 1/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 1/12 | 0/12 — Any report of weakness 1 hour following the meal (after the clamp procedure).
Hungry-during past week (General disorders) | 10/14 | 12/14 | 5/5 | 4/5 | 5/6 | 5/6 | 9/12 | 8/12 — Any report of hunger anytime during the past 7 days.
Hungry-prior to injection (General disorders) | 11/14 | 11/14 | 5/5 | 5/5 | 5/6 | 4/5 | 9/12 | 8/12 — Any report of hunger prior to injection of antipsychotic or saline.
Hungry-30 minutes post injection (General disorders) | 10/14 | 11/14 | 5/5 | 5/5 | 6/6 | 5/6 | 10/12 | 10/12 — Any report of hunger 30 minutes following an injection of antipsychotic or saline.
Hungry-end of clamp (General disorders) | 8/14 | 9/14 | 4/5 | 4/5 | 5/6 | 4/6 | 7/12 | 9/12 — Any report of hunger at the end of the clamp procedure.
Hungry-1 hour post meal (General disorders) | 0/14 | 0/14 | 1/5 | 0/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of hunger 1 hour following the meal (after the clamp procedure).
Pain-during past week (General disorders) | 2/14 | 2/14 | 0/5 | 2/5 | 0/6 | 1/6 | 1/12 | 1/12 — Any report of pain anytime during the past 7 days.
Pain-prior to injection (General disorders) | 0/14 | 4/14 | 0/5 | 0/5 | 1/6 | 1/6 | 0/12 | 2/12 — Any report of pain prior to injection of antipsychotic or saline.
Pain-30 minutes post injection (General disorders) | 0/14 | 3/14 | 0/5 | 0/5 | 0/6 | 2/6 | 1/12 | 1/12 — Any report of pain 30 minutes following an injection of antipsychotic or saline.
Pain-end of clamp (General disorders) | 0/14 | 2/14 | 0/5 | 0/5 | 0/6 | 1/6 | 0/12 | 0/12 — Any report of pain at the end of the clamp procedure.
Pain-1 hour post meal (General disorders) | 1/14 | 2/14 | 0/5 | 0/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of pain 1 hour following the meal (after the clamp procedure).
Other-Neck uncomfortable (end of clamp) (General disorders) | 1/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 0/12 | 0/12 — Other-neck uncomfortable, "pillow too big" at the end of the clamp procedure.
Other-Neck uncomfortable (1 hour post meal) (General disorders) | 1/14 | 0/14 | 0/5 | 0/5 | 0/6 | 0/6 | 0/12 | 0/12 — Other-neck uncomfortable, "pillow too big" 1 hour following the meal (after the clamp procedure).
Dizziness-end of clamp (General disorders) | 0/14 | 0/14 | 0/5 | 1/5 | 0/6 | 0/6 | 0/12 | 0/12 — Any report of dizziness at the end of the clamp procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No